CLINICAL TRIAL: NCT00314418
Title: Patient Position and Impact on Colonoscopic Cecal Intubation Time
Brief Title: Patient Position and Impact on Colonoscopy Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SV0001; Digestive Disease
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2006-04-13 (Estimated); Status verified 2006-04

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; technique; time; duration; position; abdominal pressure
MeSH Terms: interventions — Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy in the prone position

SUMMARY:
Colonoscopy is usually associated with coiling ("looping") of the colonoscope (instrument used for the procedure) in parts of the bowel. This is the main reason for patient discomfort and lengthens the duration of the procedure. Minimizing the coiling of the colonoscope would decrease the duration, and improve the efficiency and tolerability of the procedure and have a positive impact on colon cancer screening.

The primary aim of this study is to compare the time it takes for the colonoscope to reach the end of the colon when the patient is lying on the belly versus the left side (usual) at the start of the procedure. Patients who have medical conditions that may be affected by lying on their belly or those who cannot comfortably lie on the belly will be excluded from the study. Changes in patient position and use of abdominal pressure (commonly given by the endoscopy nurse during the procedure) will be permitted as necessary and determined by the endoscopist. The endoscopist will also retain the decision to discontinue the patient's participation from the study for any medical reason. After the procedure the patient will be monitored in the usual manner and asked to fill out a "satisfaction survey" (24 hours after).

DETAILED DESCRIPTION:
1. Principal investigator: Shivakumar Vignesh MD, Gastroenterology Attending Physician, VACHS

Colonoscopy with the patient in the prone position may reduce colonoscopy duration and may reduce patient discomfort by a reduction in coiling of the colonoscope with a mobile part of the bowel, decreased need for abdominal pressure and less sedation may improve the safety and efficacy of colonoscopy.

Objective: To determine if starting colonoscopy with the patient in the prone position will reduce cecal intubation time (time to reach the cecum) and total sedation requirement.

Subjects: 120 adult male, patients referred of outpatient colonoscopy will be the study subjects and controls. We do 15-18 colonoscopies a day and assuming half that number meet criteria for inclusion and consent to the study we will be able to recruit 120 patients in 6 months or less. Our records indicate more than 1000 colonoscopies are performed in a six-month period. If we conservatively estimate 10% ineligible patients > (n=900 remaining), 50% refusal (n=450 remaining), and enrollment on 4 of 5 weekdays (n=360 remaining), the six-month period would provide adequate sample size. The study would end if the target sample size is reached early.

Inclusion criteria: All adult, male patients presenting for outpatient colonoscopy. Patients who have had colonoscopies in the past and those who present for their first colonoscopy will be invited to participate in the study. It will not matter if it is their first or repeat colonoscopy as they will be randomized to either position.

Exclusion criteria: Severe obstructive lung disease requiring home oxygen, congestive heart failure not adequately managed, other conditions causing breathing difficulty, massive ascites (fluid accumulation causing a tensely distended abdomen), or inability to lie prone for any reason. Patients allergic to Versed or Fentanyl will be excluded from the study.

All female patients will be excluded as they comprise less than 2% of our colonoscopies and we don't routinely check if female patients are pregnant and the safety of lying prone during colonoscopy in pregnancy is unknown.

No vulnerable population(s) will be included.

Selection: At the time of presentation for outpatient colonoscopy, patients satisfying the inclusion and exclusion criteria will be educated about the purpose, risks and benefits of the study and informed consent will be obtained.

Participants will be randomized using a permuted block scheme with equal allocation among treatment arms. Treatment will be initiated immediately following random assignment.

The statistician will release the randomization scheme and assignments to Karl Larson PA (not involved in the study) who will inform the PI of the study assignment after patients are consented, prior to the colonoscopy.

Recruitment: For our single center (VACHS) study we plan to enroll a total of 120 patients among the patients presenting for outpatient colonoscopy, 60 in each arm. Dr.Vignesh (PI) will select patients by applying the inclusion and exclusion criteria, review their VA medical record, take a history and a physical (done before every colonoscopy) and at the same time will obtain the consent for both the colonoscopy and the study. They will be randomized using a permuted block randomization scheme and allocation concealed till the start of procedure.

Research Plan: Single-center (VACHS), Prospective, randomized, controlled, non-blinded (The GI fellow doing the data analysis, will be blinded to the assignment) study of positioning for colonoscopy in veterans undergoing outpatient colonoscopy.

Basis of sample size calculation: The national average time for cecal intubation is 15 minutes. A reduction in the colonoscopy duration by 3 minutes would be clinically meaningful and reduce cost. We do 15-20 outpatient colonoscopies in two rooms with one nurse per room daily at the West Haven VA and a reduction of 3 minutes per colonoscopy will save 45-60 minutes per day and this does not include the potential reduction in recovery time from using less sedation.

Sample size calculations, using nQuery Advisor, assuming 15 minutes for a standard procedure, and 12 minutes for a prone procedure (common standard > deviation of 5 minutes); the difference in duration of 2 minutes has important public health implications and was considered clinically meaningful in other studies of modifications in Colonoscopy procedures (4,5,6,7,8,9). Using a two-tail alpha error of 0.05, and beta error of 0.10 (power >90% ), 60 patients in each arm would be required (120 total). The study would end if the target sample size is reached early.

Methodology:

The bowel preparation, type of colonoscopes, techniques (including polypectomy) will be the same as our routine practice, they are mentioned below to be complete.

All patients who undergo outpatient colonoscopy at our institution receive the following as bowel preparation:

1. Clear liquid diet 24 hours prior to procedure
2. One gallon of Golytely the day prior to colonoscopy starting at noon.
3. Patients with serum creatinine under 2.0 to drink 300 cc of magnesium citrate following the Golytely.

Standard adult colonoscopes only will be used. Polyps will be removed with snare polypectomy or biopsy upon withdrawal of the colonoscope from the cecum as is the normal practice. In the event of failure to reach the cecum with the standard adult colonoscope, a variable-stiffness colonoscope (adult or pediatric) will be used (4, 6). In patients with severe stenosing diverticular disease, with difficulty in navigating the affected segment a pediatric variable stiffness colonoscope will be used (5).

Midazolam and Fentanyl will be the only medications used, their doses depending on the patient's vital signs and discomfort.

Vital signs will be monitored every 5 minutes during the procedure. All patients will be placed on oxygen 2 liters via nasal cannula prior to commencement of colonoscopy.

After starting the procedure changes in patient's position or abdominal pressure will be documented.

Baseline data and demographic information including height, weight, age, co-morbid illnesses and history of abdominal surgery will be collected from each patient to enable comparison between the two arms.

After starting the procedure if the patient's position is altered or abdominal pressure is used to help with the colonoscopy it will be documented as "position change" and "abdominal pressure" but there will be no crossover. Our study is not powered to measure differences between "position changes" or "abdominal pressure" these will merely be described. The patients whose position is altered will be analyzed based on the original group assignment (Intent to treat analysis).

Complications of colonoscopy being rare (Bleeding < 1%) and perforation (< 0.02%) will be described if they occur but our study is not powered to analyze them.

Primary Endpoint:

1) Time to cecal intubation

Secondary Endpoint:

1) Total medication (Midazolam and Fentanyl) dose dichotomized to low ( Midazolam 4mg IV or less, Fentanyl 200 mcg IV or less) or high (Midazolam> 4 mg IV and Fentanyl >200 mcg IV).

The time to cecal intubation will be measured and a t-test will be used to compare the difference between the mean duration.

The total opiate doses will be recorded and dichotomized to low ( Midazolam 4mg IV or less, Fentanyl 200 mcg IV or less) or high (Midazolam> 4 mg IV and Fentanyl >200 mcg IV) compared using the Chi-square test.

The prone position (lying on the belly) does not increase risk of complications based on our experience. We have done hundreds of colonoscopies safely in the prone position. The prone position with the patient's head turned to one side may reduce aspiration risk as it facilitates the drainage of secretions via the mouth. By applying our exclusion criteria we do not offer the study to a patient with a medical condition that is affected by lying on the belly.

Colonoscopies are done with "conscious sedation", last 30 minutes and have the same stringent cardio respiratory monitoring. For this study we will follow our standard continuous cardio-respiratory monitoring, blood pressure measurements every 5 minutes. We also administer Oxygen 2 liters by nasal cannula routinely. We have an adverse event form to document any cases of cardio-respiratory depression or any other adverse event in a procedure involving conscious sedation. The physicians involved in conscious sedation have been certified in a "Conscious sedation and airway management" course conducted by Yale New Haven hospital.

Informed Consent will be obtained for the colonoscopy outlining the risks and separately for study using the VA research consent form. The consents will be obtained in the ambulatory procedure unit after the patients are prepared for the colonoscopy.

We strictly adhere to HIPAA regulations in our daily practice. The information obtained in the study and the patient's medical record will be de-identified and accessible to the investigators mentioned above exclusively.

Your research records will be kept as confidential as possible and only the gastroenterologists and the endoscopy nurses participating in your case will have access to the information obtained for the study. Only a code number will identify your research records. The code number will not be based on any information that could be used to identify you. The master list linking names to code numbers will be kept separately from the research data. All research information will be kept in locked files at all times. Only authorized research staff will have access to the information gathered in this study. A note describing your participation in this research study will be placed in your VA medical record.

ELIGIBILITY:
Inclusion Criteria: Male Veterans presenting for outpatient colonoscopy for any indication.

Exclusion Criteria:

* Severe Congestive heart failure with left Ventricular ejection fraction <30%,
* Severe Chronic Obstructive lung disease dependant on Home Oxygen or recent decompensation,
* Spine disease or other condition with difficulty laying in the prone position.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09; Study Completion 2006-03

PRIMARY OUTCOMES:
Colonoscopic Cecal Intubation time

SECONDARY OUTCOMES:
Total colonoscopy time, colonoscope withdrawal time, cumulative sedation dose, recovery time, need for abdominal pressure and changes in patient position during the procedure, adenoma prevalence rate, complications, patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Shivakumar Vignesh, MD, Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States